CLINICAL TRIAL: NCT04202094
Title: Follow-up of Fertility in Young Adults Who Did or Did Not Store Testicular Tissue Before Gonadotoxic Treatment for Fertility Preservation
Brief Title: Fertility in Young Adults Who Did (Not) Store Testicular Tissue Before a Treatment Leading to Fertility Problems
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Ellen Goossens, Head of research group BITE, Vrije Universiteit Brussel
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-342
Record Dates: First submitted 2019-12-06; First posted 2019-12-17 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Childhood Cancer; Hematological Disorders
Keywords: Male fertility preservation; Testicular tissue biopsy; Male fertility status; Tanner stage; Testicular volume; Hormones; Semen analysis
MeSH Terms: conditions — Neoplasms; Hematologic Diseases | interventions — Physical Examination; Blood Specimen Collection; Semen Analysis

STUDY DESIGN:
Intervention Model Description: This study is a prospective comparative interventional cohort study.
  The fertility status of young adults (≥18 years) cured of childhood cancer or hematological disorders for which they received high-risk gonadotoxic treatment (with an ≥80% risk of later fertility problems) during childhood will be compared between patients who did and those who did not undergo a testicular tissue biopsy procedure at a young age as a fertility preservation strategy in order to identify a possible association between the biopsy procedure (which is performed to harvest testicular tissue) and the later fertility outcome.
  Their fertility status will also be compared to the reproductive health of spontaneously conceived young adults that has already been published (Belva F et al., 2016/2017/2019).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Biopsy group (Experimental): Young adult men (≥18 years) cured of childhood cancer or hematological disorders for which they received high-risk gonadotoxic treatment during childhood and who have chosen to undergo a testicular biopsy procedure at a young age as a fertility preservation strategy.
  Interventions: Diagnostic Test: Physical examination; Diagnostic Test: Scrotum ultrasound; Diagnostic Test: Blood sample; Diagnostic Test: Semen analysis
- No biopsy group (Experimental): Young adult men (≥18 years) cured of childhood cancer or hematological disorders for which they received high-risk gonadotoxic treatment during childhood and who have refused to undergo a testicular biopsy procedure at a young age as a fertility preservation strategy.
  Interventions: Diagnostic Test: Physical examination; Diagnostic Test: Scrotum ultrasound; Diagnostic Test: Blood sample; Diagnostic Test: Semen analysis
- Control group (No Intervention): Spontaneously conceived young adults whose data on reproductive health have already been published (Belva F et al., 2016/2017/2019).

INTERVENTIONS:
Diagnostic Test: Physical examination — A physical examination to measure the patients' weight, height, body mass index, blood pressure and testicular volume using a Prader orchidometer and to determine the patients' Tanner stage (secondary sexual development).
  Arms: Biopsy group; No biopsy group
Diagnostic Test: Scrotum ultrasound — A scrotum ultrasound to measure the patients' testicular volume and to investigate potential abnormalities in the testicular parenchyma.
  Arms: Biopsy group; No biopsy group
Diagnostic Test: Blood sample — A morning blood sample to evaluate the serum levels of luteinizing hormone (LH), follicle-stimulating hormone (FSH), testosterone (T), estradiol (E2), inhibin B (INHB), thyroid-stimulating hormone (TSH), free thyroxine (FT4), insulin-like growth factor 1 (IGF1), prolactin (PRL), cortisol and adrenocorticotropic hormone (ACTH). Upon approval by the patient himself, a spare blood sample will be collected and retained for 5 years for subsequent research purposes limited to the context of the present study.
  Arms: Biopsy group; No biopsy group
Diagnostic Test: Semen analysis — A semen analysis to evaluate ejaculate volume, sperm concentration, sperm motility, and sperm morphology. If sperm is found in the semen sample, an anti-sperm antibody test and a sperm DNA fragmentation test will be performed. Upon approval by the patient himself, the surplus of the semen sample will be retained for 5 years for subsequent research purposes limited to the context of the present study.
  Arms: Biopsy group; No biopsy group

SUMMARY:
The goal of this prospective comparative interventional cohort study is to assess the fertility status of young adult men (≥18 years) who received gonadotoxic treatment during childhood for the treatment of cancer or hematological disorders. These treatment protocols are highly gonadotoxic (i.e. they may cause later fertility problems) and therefore these patients have been proposed to store some testicular tissue during childhood as an option to preserve their fertility.

The main questions this study aims to answer are (1) the impact of the received gonadotoxic treatment on the later fertility status and (2) the additional impact of a testicular biopsy procedure (performed at a young age to harvest testicular tissue for storage) on the future fertility.

Participants will be asked to undergo a physical examination by a fertility specialist, to undergo a scrotal ultrasound, to give a blood sample, and to provide a semen sample.

Researchers will compare the patients fertility status between the different received gonadotoxic treatment protocols, between patients who underwent a testicular biopsy procedure at a young age and those who did not, and compare the patients fertility status with the reproductive health of spontaneously conceived young adults.

DETAILED DESCRIPTION:
See the subsequent protocol sections.

ELIGIBILITY:
Inclusion criteria

* young adult men (≥18 years)
* diagnosis of cancer or hematological disorder during childhood (<18 years)
* high-risk gonadotoxic treatment received during childhood
* at least one year after the last received genotoxic treatment
* did/did not undergo a testicular biopsy procedure at a young age for fertility preservation

Exclusion criteria

- prepubertal patients and adolescents (<18 years)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Impact of childhood gonadotoxic treatment on fertility status | at baseline and in 1 year
  The patients' fertility status (physical examination, scrotum ultrasound, blood sample, semen analysis) will be evaluated once a year after cessation of the gonadotoxic treatment. Only in case of infertility (azoospermia) or subfertility (oligo-, astheno- or teratozoospermia), the different interventions will be repeated one year later as the recovery of spermatogenesis with return of sperm production may occur several years after gonadotoxic treatment.

SECONDARY OUTCOMES:
Impact of testicular biopsy procedure (performed at a young age) on fertility status | at baseline and in 1 year
  The patients' fertility status (physical examination, scrotum ultrasound, blood sample, semen analysis) will be evaluated once a year after cessation of the gonadotoxic treatment. Only in case of infertility (azoospermia) or subfertility (oligo-, astheno- or teratozoospermia), the different interventions will be repeated one year later as the recovery of spermatogenesis with return of sperm production may occur several years after gonadotoxic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Goossens, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delgouffe E, Braye A, Vloeberghs V, Mateizel I, Ernst C, Ferster A, Devalck C, Tournaye H, Gies I, Goossens E. Spermatogenesis after gonadotoxic childhood treatment: follow-up of 12 patients. Hum Reprod Open. 2023 Jul 31;2023(3):hoad029. doi: 10.1093/hropen/hoad029. eCollection 2023. PMID 37547664
- [Background] Belva F, Bonduelle M, Roelants M, Michielsen D, Van Steirteghem A, Verheyen G, Tournaye H. Semen quality of young adult ICSI offspring: the first results. Hum Reprod. 2016 Dec;31(12):2811-2820. doi: 10.1093/humrep/dew245. Epub 2016 Oct 5. PMID 27707840
- [Background] Belva F, Roelants M, De Schepper J, Van Steirteghem A, Tournaye H, Bonduelle M. Reproductive hormones of ICSI-conceived young adult men: the first results. Hum Reprod. 2017 Feb;32(2):439-446. doi: 10.1093/humrep/dew324. Epub 2016 Dec 21. PMID 28007789
- [Background] Belva F, Bonduelle M, Tournaye H. Endocrine and reproductive profile of boys and young adults conceived after ICSI. Curr Opin Obstet Gynecol. 2019 Jun;31(3):163-169. doi: 10.1097/GCO.0000000000000538. PMID 30870183